CLINICAL TRIAL: NCT04463823
Title: Covid-19 Convalescent Plasma Used for Treatment of Patients in Norway - a Monitoring Study
Brief Title: "NORPLASMA" Covid-19 Convalescent Plasma Treatment Monitoring Study
Acronym: MONITOR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset Telemark (Other Government); Sykehuset Ostfold (Other); University Hospital, Akershus (Other); Sorlandet Hospital HF (Other Government); Helse Fonna (Other)
Responsible Party: Principal Investigator, Lise Sofie Haug Nissen-Meyer, Project manager, Oslo University Hospital
Other Study IDs: 148622
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: COVID
Keywords: Convalescent plasma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NORPLASMA COVID-19 includes both the production of convalescent plasma from approved blood donors who have recovered from covid-19 (coronavirus disease 2019), and clinical studies to evaluate efficacy and safety of the treatment, as recommended by European health authorities. Patients who receive convalescent plasma in a clinical setting will be invited to participate in the monitoring study NORPLASMA MONITOR, where clinical data about safety and effect on clinical parameters including virus load and recovery time will be collected and compared to european patients in a common database for the European countries. The treated patients can be compared to a historical control group.

DETAILED DESCRIPTION:
The NORPLASMA MONITOR study:

Main hypothesis: Plasma from selected COVID-19 convalescent blood donors contain neutralizing/therapeutic antibodies against Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) that may prevent generalized spreading of the infection if administered in a sufficient dose at the right time.

The aim of the monitoring study is to monitor the treatment, characterize antibody properties, dose requirements and safety issues.

In the NORPLASMA MONITOR study, the investigators will collect data from all patients treated with convalescent plasma in Norwegian hospitals/care institutions. The data will be compared to historical controls to evaluate efficacy, and for all transfusions, antibody characteristics and effective doses can be retrospectively calculated.

The complete protocol is available on our web site https://www.ous-research.no/home/norplasma.

Patients receiving COVID-19 convalescent plasma on a clinical indication as part of their treatment should be included in the MONITOR study.

The purpose of the monitoring study is to collect as much clinical information as possible about patients with COVID-19 before and after administration of convalescent plasma, together with extensive data about blood donors and their antibody properties. Because the plasma units cannot be fully standardized before use, it is of vital importance to record enough data to allow necessary analysis and calculations, of e.g., antibody concentration in each recipient. Data will also be shared within the European Union (EU) to obtain results in a more efficient way from larger materials.

For the execution of this study, the project group intends to establish cooperation with all hospitals/care institutions with transfusion procedures where COVID-19-patients are treated. Contact will be established via local coordinators in the blood centers, and clinical cooperation partners in relevant hospital departments will be recruited consecutively as COVID-19 patients where plasma treatment is considered indicated, are admitted. Since the treatment will be offered to these patients independent of study inclusion, it is important to communicate the value of the patient inclusion and data collection to their responsible care providers, so that participation can be encouraged.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with covid-19 convalescent plasma
* patients who has provided informed consent or where nearest relative has given consent

Exclusion Criteria:

* patients included in other clinical studies of covid-19 treatment
* consent not given

All eligible patients should be invited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to health institutions where transfusion therapy is routinely given, and who are receiving COVID-19 convalescent plasma on a clinical indication as part of their treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
observation | up to 2 years
  clinical data and lab results from patients who receive COVID-19 convalescent plasma on a clinical indication, are being collected for later analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lise Sofie Haug Nissen-Meyer, Ph.D., Principal Investigator — Oslo University Hospital
Locations (7):
- Norway (7):
  - Helse Fonna, Haugesund
  - Sorlandet hospital, Kristiansand
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Sykehuset Ostfold, Sarpsborg
  - Sykehuset Telemark, Skien
  - St.Olavs Hospital, Trondheim